CLINICAL TRIAL: NCT00821561
Title: A Phase 2, Randomized, Prospective, Double-masked, Vehicle-controlled, Dose-ranging Study to Evaluate the Efficacy and Safety of Nexagon® in Subjects With Persistent Corneal Epithelial Defects (PED) From Chemical Burn Injuries.
Brief Title: A Study to Investigate the Safety and Clinical Effect of Nexagon® to Treat Persistent Epithelial Defects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn prior to recruitment for business reasons.
Sponsor: OcuNexus Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEX-PED-001
Record Dates: First submitted 2009-01-10; First posted 2009-01-13 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: Persistent Epithelial Defect
Keywords: Persistent; cornea; defect; Nexagon; Coda
MeSH Terms: conditions — Corneal Diseases; Cavitary Optic Disc Anomalies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nexagon®
Drug: Nexagon® vehicle

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Nexagon® in subjects with Persistent Epithelial Defects (PED) originally caused by chemical burns.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 years and over.
2. Subjects who are able to attend all follow-up visits and who are able to comply with all study procedures.
3. Subjects who are willing and able to give written informed consent to take part in the study.
4. At the Day -7 visit subjects must have a corneal epithelial defect that has persisted for between 7 days and 14 days, which has a minimum diameter of 2 mm along the greatest axis, and which has not shown improvement despite conventional treatment such as tear supplements and bandage contact lenses.
5. The original defect to the cornea must have been caused by either alkaline or acidic agents.

Exclusion Criteria:

1. Use of concomitant ocular medications in the screening period that are not specified in standardized PED treatment regime
2. Likely to require the use of concomitant ocular medications that are not specified in the standardized PED treatment regime during the study follow-up period
3. Decrease or increase in the PED by more than 30% during the screening period.
4. Have an active lid or ocular infectious process of any sort
5. Subjects with corneal perforation or impending corneal perforation
6. The circumference affected by limbal blood vessel ischemia is greater than 75% of the circumference
7. Subjects with severe lid abnormalities contributory to the persistence of the PED such as inability to close the lids.
8. Subjects with bilateral PED, if the smaller PED has a longest diameter of > 2 mm.
9. Female subjects who are pregnant or breastfeeding. F
10. Subjects who have a history of AIDS or HIV.
11. Subjects with any other condition which, in the Investigator's opinion, would exclude the subject from participating.
12. Treatment with systemic corticosteroids (equivalent to > 10 mg/day of prednisone) or immunosuppressive or chemotherapeutic agents within 7 days prior to Day 0, or likely to receive one of these therapies during study participation
13. Subjects who have participated in a clinical trial within 30 days prior to Day 0.
14. Diabetics with an HbA1c greater than 6.5%.
15. Diabetics who are currently prescribed more than one oral medication for their diabetes.
16. Subjects who have more than one distinct PED in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-11 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the efficacy and safety of Nexagon® as a treatment for PED from chemical burn injuries.